CLINICAL TRIAL: NCT01077258
Title: Effectiveness and Safety of Adalimumab in Patients With Rheumatoid Arthritis in Routine Clinical Practice
Brief Title: Efficacy and Safety of Adalimumab in Patients With Rheumatoid Arthritis in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-448
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Safety; Long-term observation; Routine Clinical Setting; Rheumatoid Arthritis; Effectiveness
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis: Participants with rheumatoid arthritis prescribed adalimumab in routine clinical practice were observed from the first dose for up to 24 months.

SUMMARY:
Observation of safety, tolerability and effectiveness of adalimumab (Humira) therapy in a large patient collective under everyday clinical conditions over 2 years.

DETAILED DESCRIPTION:
Patients with rheumatoid arthritis who started treatment with adalimumab in a normal clinical setting according to the product label were documented. The follow-up observation period was for 2 years and focused on safety information and maintenance of efficacy during a normal clinical setting. Follow-up with participants was via regular office visits at intervals as determined by routine clinical practice or as recommended by national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active rheumatoid arthritis in adults with insufficient response to disease-modifying antirheumatic drugs, including methotrexate
* Moderate to severe active rheumatoid arthritis in adults who have not been treated with methotrexate before. In case of incompatibility with methotrexate, Humira can be used as monotherapy

Exclusion Criteria:

* Hypersensitivity against the drug or one of the other ingredients
* Active tuberculosis or other severe infections (e.g. sepsis and opportunistic infections)
* Moderate to severe cardiac insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample: patients with rheumatoid arthritis who resided in Germany. German regulations state that all patients are eligible for non-interventional studies; there are no exclusions. Adult patients (≥ 18 years of age) with RA who were preparing to initiate adalimumab therapy according to the product label were eligible for study enrollment. The eligibility criteria below reflect the approved label as stated in the German Summary of Product Characteristics (SPC) for Humira.
Sampling Method: Non-Probability Sample
Enrollment: 4208 (Actual)
Dates: Start 2004-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Wittig, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department
Locations (303):
- Germany (303):
  - Site Reference ID/Investigator# 35036, Aachen
  - Site Reference ID/Investigator# 35510, Ahlen
  - Site Reference ID/Investigator# 35040, Ahrensburg
  - Site Reference ID/Investigator# 35043, Altenburg
  - Site Reference ID/Investigator# 35046, Altenholz
  - Site Reference ID/Investigator# 35049, Amberg
  - Site Reference ID/Investigator# 35057, Arnstadt
  - Site Reference ID/Investigator# 35520, Attendorn
  - Site Reference ID/Investigator# 33349, Augsburg
  - Site Reference ID/Investigator# 33358, Bad Abbach
  - Site Reference ID/Investigator# 33361, Bad Abbach
  - Site Reference ID/Investigator# 35142, Bad Aibling
  - Site Reference ID/Investigator# 35570, Bad Brambach
  - Site Reference ID/Investigator# 35573, Bad Bramstedt
  - Site Reference ID/Investigator# 33372, Bad Endbach
  - Site Reference ID/Investigator# 33378, Bad Iburg
  - Site Reference ID/Investigator# 33382, Bad Iburg
  - Site Reference ID/Investigator# 33387, Bad Kreuznach
  - Site Reference ID/Investigator# 35575, Bad Kreuznach
  - Site Reference ID/Investigator# 33391, Bad Liebenwerda
  - Site Reference ID/Investigator# 33396, Bad Münder am Deister
  - Site Reference ID/Investigator# 102216, Bad Nauheim
  - Site Reference ID/Investigator# 35578, Bad Neuenahr
  - Site Reference ID/Investigator# 33404, Bad Rappenau
  - Site Reference ID/Investigator# 51883, Bad Salzungen
  - Site Reference ID/Investigator# 33412, Bad Soden-Salmünster
  - Site Reference ID/Investigator# 33425, Baden-Baden
  - Site Reference ID/Investigator# 33429, Bamberg
  - Site Reference ID/Investigator# 33438, Bautzen
  - Site Reference ID/Investigator# 33442, Bayreuth
  - Site Reference ID/Investigator# 33446, Bayreuth
  - Site Reference ID/Investigator# 33641, Berlin
  - Site Reference ID/Investigator# 35089, Berlin
  - Site Reference ID/Investigator# 33648, Berlin
  - Site Reference ID/Investigator# 33693, Berlin
  - Site Reference ID/Investigator# 33670, Berlin
  - Site Reference ID/Investigator# 33658, Berlin
  - Site Reference ID/Investigator# 33697, Berlin
  - Site Reference ID/Investigator# 34246, Berlin
  - Site Reference ID/Investigator# 33683, Berlin
  - Site Reference ID/Investigator# 34269, Berlin
  - Site Reference ID/Investigator# 35527, Berlin
  - Site Reference ID/Investigator# 35597, Berlin
  - Site Reference ID/Investigator# 33620, Berlin
  - Site Reference ID/Investigator# 33690, Berlin
  - Site Reference ID/Investigator# 33704, Berlin
  - Site Reference ID/Investigator# 33687, Berlin
  - Site Reference ID/Investigator# 33661, Berlin
  - Site Reference ID/Investigator# 35550, Berlin
  - Site Reference ID/Investigator# 33674, Berlin
  - Site Reference ID/Investigator# 35551, Berlin
  - Site Reference ID/Investigator# 34238, Berlin
  - Site Reference ID/Investigator# 35556, Bernau
  - Site Reference ID/Investigator# 34277, Biberach
  - Site Reference ID/Investigator# 35562, Binzen
  - Site Reference ID/Investigator# 34285, Blankenburg/Hart
  - Site Reference ID/Investigator# 34288, Blaubeuren Abbey
  - Site Reference ID/Investigator# 34291, Bocholt
  - Site Reference ID/Investigator# 35566, Bocholt
  - Site Reference ID/Investigator# 35641, Bochum
  - Site Reference ID/Investigator# 35644, Bogen
  - Site Reference ID/Investigator# 34302, Bonn
  - Site Reference ID/Investigator# 35646, Bonn
  - Site Reference ID/Investigator# 34296, Bonn
  - Site Reference ID/Investigator# 35652, Bottrop
  - Site Reference ID/Investigator# 34307, Braunschweig
  - Site Reference ID/Investigator# 35603, Breitenbrunn
  - Site Reference ID/Investigator# 35609, Bremen
  - Site Reference ID/Investigator# 34266, Buch
  - Site Reference ID/Investigator# 35611, Celle
  - Site Reference ID/Investigator# 34699, Chemnitz
  - Site Reference ID/Investigator# 35093, Chemnitz
  - Site Reference ID/Investigator# 35615, Coesfeld
  - Site Reference ID/Investigator# 33989, Cologne
  - Site Reference ID/Investigator# 35237, Cologne
  - Site Reference ID/Investigator# 34708, Cottbus
  - Site Reference ID/Investigator# 34711, Cottbus
  - Site Reference ID/Investigator# 35621, Darmstadt
  - Site Reference ID/Investigator# 34725, Deggendorf
  - Site Reference ID/Investigator# 35631, Dessau
  - Site Reference ID/Investigator# 34742, Dortmund
  - Site Reference ID/Investigator# 35635, Dortmund
  - Site Reference ID/Investigator# 35634, Dortmund
  - Site Reference ID/Investigator# 35170, Dresden
  - Site Reference ID/Investigator# 34754, Dresden
  - Site Reference ID/Investigator# 34748, Dresden
  - Site Reference ID/Investigator# 34751, Dresden
  - Site Reference ID/Investigator# 34760, Dresden
  - Site Reference ID/Investigator# 34778, Duisburg
  - Site Reference ID/Investigator# 34773, Düsseldorf
  - Site Reference ID/Investigator# 34768, Düsseldorf
  - Site Reference ID/Investigator# 34784, Eberswalde
  - Site Reference ID/Investigator# 35184, Elmshorn
  - Site Reference ID/Investigator# 34809, Erfurt
  - Site Reference ID/Investigator# 35096, Erfurt
  - Site Reference ID/Investigator# 35191, Erfurt
  - Site Reference ID/Investigator# 34821, Erlangen
  - Site Reference ID/Investigator# 35196, Essen
  - Site Reference ID/Investigator# 35199, Essen
  - Site Reference ID/Investigator# 35202, Feldafing
  - Site Reference ID/Investigator# 35205, Flensburg
  - Site Reference ID/Investigator# 34833, Forchheim
  - Site Reference ID/Investigator# 35210, Frankenberg
  - Site Reference ID/Investigator# 34849, Frankfurt
  - Site Reference ID/Investigator# 34840, Frankfurt
  - Site Reference ID/Investigator# 34843, Frankfurt
  - Site Reference ID/Investigator# 35213, Fraureuth
  - Site Reference ID/Investigator# 35219, Freiberg
  - Site Reference ID/Investigator# 34854, Freiburg im Breisgau
  - Site Reference ID/Investigator# 35221, Freiburg im Breisgau
  - Site Reference ID/Investigator# 34861, Freiburg im Breisgau
  - Site Reference ID/Investigator# 35101, Freystadt
  - Site Reference ID/Investigator# 35224, Friedrichroda
  - Site Reference ID/Investigator# 34879, Gelsenkirchen
  - Site Reference ID/Investigator# 34883, Gera
  - Site Reference ID/Investigator# 34887, Giessen
  - Site Reference ID/Investigator# 35491, Gosheim
  - Site Reference ID/Investigator# 34896, Goslar
  - Site Reference ID/Investigator# 34901, Greifswald
  - Site Reference ID/Investigator# 35496, Greifswald
  - Site Reference ID/Investigator# 34904, Greifswald
  - Site Reference ID/Investigator# 102217, Groß Ammensleben
  - Site Reference ID/Investigator# 33897, Groß Reken
  - Site Reference ID/Investigator# 35498, Guben
  - Site Reference ID/Investigator# 34912, Güstrow
  - Site Reference ID/Investigator# 35503, Hagen
  - Site Reference ID/Investigator# 34937, Halle
  - Site Reference ID/Investigator# 34940, Halle
  - Site Reference ID/Investigator# 34922, Halle
  - Site Reference ID/Investigator# 34944, Halle
  - Site Reference ID/Investigator# 34932, Halle
  - Site Reference ID/Investigator# 35444, Hamburg
  - Site Reference ID/Investigator# 35441, Hamburg
  - Site Reference ID/Investigator# 34970, Hamburg
  - Site Reference ID/Investigator# 34952, Hamburg
  - Site Reference ID/Investigator# 34958, Hamburg
  - Site Reference ID/Investigator# 35452, Hamburg
  - Site Reference ID/Investigator# 35007, Hamburg
  - Site Reference ID/Investigator# 35000, Hamburg
  - Site Reference ID/Investigator# 34961, Hamburg
  - Site Reference ID/Investigator# 35449, Hamburg
  - Site Reference ID/Investigator# 34955, Hamburg
  - Site Reference ID/Investigator# 34998, Hamburg
  - Site Reference ID/Investigator# 34994, Hamburg
  - Site Reference ID/Investigator# 34983, Hamburg
  - Site Reference ID/Investigator# 34986, Hamburg
  - Site Reference ID/Investigator# 35111, Hamburg
  - Site Reference ID/Investigator# 34974, Hamburg
  - Site Reference ID/Investigator# 35019, Hanau
  - Site Reference ID/Investigator# 33712, Hanover
  - Site Reference ID/Investigator# 35025, Hanover
  - Site Reference ID/Investigator# 33792, Harrislee
  - Site Reference ID/Investigator# 35459, Haselünne
  - Site Reference ID/Investigator# 102215, Heidelberg
  - Site Reference ID/Investigator# 33798, Heidelberg
  - Site Reference ID/Investigator# 35119, Heidelberg
  - Site Reference ID/Investigator# 33801, Heidelberg
  - Site Reference ID/Investigator# 33808, Heidelberg
  - Site Reference ID/Investigator# 35464, Heidenheim
  - Site Reference ID/Investigator# 33818, Heilbad Heiligenstadt
  - Site Reference ID/Investigator# 33825, Herrsching am Ammersee
  - Site Reference ID/Investigator# 33834, Hof
  - Site Reference ID/Investigator# 33842, Hofheim
  - Site Reference ID/Investigator# 33845, Hohenfelde
  - Site Reference ID/Investigator# 33855, Illertissen
  - Site Reference ID/Investigator# 33858, Immenstadt im Allgäu
  - Site Reference ID/Investigator# 35479, Ingolstadt
  - Site Reference ID/Investigator# 51882, Jena
  - Site Reference ID/Investigator# 33942, Jülich
  - Site Reference ID/Investigator# 33946, Kahla
  - Site Reference ID/Investigator# 35125, Kahla
  - Site Reference ID/Investigator# 33950, Kaiserslautern
  - Site Reference ID/Investigator# 33956, Karlsruhe
  - Site Reference ID/Investigator# 33961, Karlsruhe
  - Site Reference ID/Investigator# 33964, Kassel
  - Site Reference ID/Investigator# 34002, Königs Wusterhausen
  - Site Reference ID/Investigator# 34008, Kressbronn
  - Site Reference ID/Investigator# 34084, Kronach
  - Site Reference ID/Investigator# 34005, Lahr
  - Site Reference ID/Investigator# 35245, Landau
  - Site Reference ID/Investigator# 34112, Leipzig
  - Site Reference ID/Investigator# 34106, Leipzig
  - Site Reference ID/Investigator# 34109, Leipzig
  - Site Reference ID/Investigator# 34100, Leipzig
  - Site Reference ID/Investigator# 35254, Lippstadt
  - Site Reference ID/Investigator# 35306, Ludwigsfelde
  - Site Reference ID/Investigator# 35262, Ludwigshafen
  - Site Reference ID/Investigator# 34136, Lübeck
  - Site Reference ID/Investigator# 34139, Lüneburg
  - Site Reference ID/Investigator# 34147, Magdeburg
  - Site Reference ID/Investigator# 34150, Magdeburg
  - Site Reference ID/Investigator# 35276, Mainz
  - Site Reference ID/Investigator# 34192, Marktredwitz
  - Site Reference ID/Investigator# 34196, Marl
  - Site Reference ID/Investigator# 34200, Meissen
  - Site Reference ID/Investigator# 35285, Menz
  - Site Reference ID/Investigator# 35287, Minden
  - Site Reference ID/Investigator# 34208, Mittelherwigsdorf
  - Site Reference ID/Investigator# 34221, Moenkeberg
  - Site Reference ID/Investigator# 34218, Mönchengladbach
  - Site Reference ID/Investigator# 34213, Mönchengladbach
  - Site Reference ID/Investigator# 34040, Munich
  - Site Reference ID/Investigator# 35295, Munich
  - Site Reference ID/Investigator# 34232, Munich
  - Site Reference ID/Investigator# 34235, Munich
  - Site Reference ID/Investigator# 35298, Munich
  - Site Reference ID/Investigator# 34043, Munich
  - Site Reference ID/Investigator# 34224, Mühlhausen
  - Site Reference ID/Investigator# 35292, Mülheim
  - Site Reference ID/Investigator# 34229, Müllheim
  - Site Reference ID/Investigator# 34048, Münster
  - Site Reference ID/Investigator# 34052, Naunhof
  - Site Reference ID/Investigator# 34061, Neubrandenburg
  - Site Reference ID/Investigator# 34064, Neuburg am Inn
  - Site Reference ID/Investigator# 34071, Neumünster
  - Site Reference ID/Investigator# 35313, Neuss
  - Site Reference ID/Investigator# 34076, Neustadt
  - Site Reference ID/Investigator# 35321, Niederbrombach
  - Site Reference ID/Investigator# 34080, Niefern-Öschelbronn
  - Site Reference ID/Investigator# 34158, Nienburg
  - Site Reference ID/Investigator# 34173, Oelsnitz
  - Site Reference ID/Investigator# 34176, Offenburg
  - Site Reference ID/Investigator# 33492, Oldenburg
  - Site Reference ID/Investigator# 34718, Ostseebad Damp
  - Site Reference ID/Investigator# 35335, Paderborn
  - Site Reference ID/Investigator# 33508, Parchim
  - Site Reference ID/Investigator# 35340, Passau
  - Site Reference ID/Investigator# 33517, Pfullendorf
  - Site Reference ID/Investigator# 67482, Pirna
  - Site Reference ID/Investigator# 33523, Planegg
  - Site Reference ID/Investigator# 33528, Plauen
  - Site Reference ID/Investigator# 33470, Potsdam
  - Site Reference ID/Investigator# 33466, Potsdam
  - Site Reference ID/Investigator# 33476, Prüm
  - Site Reference ID/Investigator# 33479, Püttlingen
  - Site Reference ID/Investigator# 33484, Radebeul
  - Site Reference ID/Investigator# 35347, Radebeul
  - Site Reference ID/Investigator# 35136, Ratingen
  - Site Reference ID/Investigator# 33488, Ratzeburg
  - Site Reference ID/Investigator# 33890, Regensburg
  - Site Reference ID/Investigator# 33883, Regensburg
  - Site Reference ID/Investigator# 33886, Regensburg
  - Site Reference ID/Investigator# 33902, Rendsburg
  - Site Reference ID/Investigator# 33907, Rheine
  - Site Reference ID/Investigator# 35355, Rickenbach
  - Site Reference ID/Investigator# 33911, Riesa
  - Site Reference ID/Investigator# 33914, Rinteln
  - Site Reference ID/Investigator# 33923, Rostock
  - Site Reference ID/Investigator# 33927, Rostock
  - Site Reference ID/Investigator# 33931, Rothenburg
  - Site Reference ID/Investigator# 35362, Rüdersdorf
  - Site Reference ID/Investigator# 34016, Saarbrücken
  - Site Reference ID/Investigator# 35383, Saint Martin
  - Site Reference ID/Investigator# 34023, Salzwedel
  - Site Reference ID/Investigator# 34027, Sande
  - Site Reference ID/Investigator# 33534, Schneeberg
  - Site Reference ID/Investigator# 33539, Schramberg
  - Site Reference ID/Investigator# 33542, Schutterwald
  - Site Reference ID/Investigator# 35371, Schwandorf in Bayern
  - Site Reference ID/Investigator# 33549, Schwerin
  - Site Reference ID/Investigator# 35376, Schwerin
  - Site Reference ID/Investigator# 33555, Schwerte
  - Site Reference ID/Investigator# 33559, Seesen
  - Site Reference ID/Investigator# 33563, Senden
  - Site Reference ID/Investigator# 35380, Singen
  - Site Reference ID/Investigator# 33567, Sinsheim
  - Site Reference ID/Investigator# 33572, Soltau
  - Site Reference ID/Investigator# 33577, Spremberg
  - Site Reference ID/Investigator# 33588, Stadthagen
  - Site Reference ID/Investigator# 33592, Steinhagen
  - Site Reference ID/Investigator# 33604, Stuttgart
  - Site Reference ID/Investigator# 33607, Stuttgart
  - Site Reference ID/Investigator# 33611, Stuttgart
  - Site Reference ID/Investigator# 33598, Stuttgart
  - Site Reference ID/Investigator# 35389, Suhl
  - Site Reference ID/Investigator# 35391, Tegernau
  - Site Reference ID/Investigator# 33625, Torgelow
  - Site Reference ID/Investigator# 33637, Ueberlingen-Nussdorf
  - Site Reference ID/Investigator# 35395, Uffenheim
  - Site Reference ID/Investigator# 33721, Ulm
  - Site Reference ID/Investigator# 33724, Ulm
  - Site Reference ID/Investigator# 33734, Viersen
  - Site Reference ID/Investigator# 33737, Villingen-Schwenningen
  - Site Reference ID/Investigator# 35397, Vöhringen
  - Site Reference ID/Investigator# 33742, Waltrop
  - Site Reference ID/Investigator# 34252, Wannsee
  - Site Reference ID/Investigator# 33749, Weener
  - Site Reference ID/Investigator# 33751, Weißenfels
  - Site Reference ID/Investigator# 33852, Welzow
  - Site Reference ID/Investigator# 35404, Wiefelstede
  - Site Reference ID/Investigator# 33761, Wiesbaden
  - Site Reference ID/Investigator# 35408, Wiesbaden
  - Site Reference ID/Investigator# 33765, Wiesbaden
  - Site Reference ID/Investigator# 35413, Wiesbaden
  - Site Reference ID/Investigator# 33772, Wilhelmshaven
  - Site Reference ID/Investigator# 33780, Wittlich
  - Site Reference ID/Investigator# 35420, Wuppertal
  - Site Reference ID/Investigator# 33718, Würzburg
  - Site Reference ID/Investigator# 33864, Zerbst
  - Site Reference ID/Investigator# 33867, Zeven
  - Site Reference ID/Investigator# 33873, Zwickau
  - Site Reference ID/Investigator# 33876, Zwickau
  - Site Reference ID/Investigator# 33880, Zwiesel

REFERENCES:
- [Derived] Behrens F, Koehm M, Schwaneck EC, Schmalzing M, Wittig BM, Gnann H, Greger G, Tony HP, Burkhardt H. Addition or removal of concomitant methotrexate alters adalimumab effectiveness in rheumatoid arthritis but not psoriatic arthritis. Scand J Rheumatol. 2019 Sep;48(5):375-382. doi: 10.1080/03009742.2019.1600717. Epub 2019 Jul 16. PMID 31311386
- [Derived] Scharbatke EC, Behrens F, Schmalzing M, Koehm M, Greger G, Gnann H, Burkhardt H, Tony HP. Association of Improvement in Pain With Therapeutic Response as Determined by Individual Improvement Criteria in Patients With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2016 Nov;68(11):1607-1615. doi: 10.1002/acr.22884. Epub 2016 Oct 1. PMID 26990995
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis: Participants with rheumatoid arthritis prescribed adalimumab in routine clinical practice were observed for up to 24 months.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis
Started | 4208
Completed | 1640
Not Completed | 2568
Not completed — Lost to Follow-up | 1390
Not completed — Adverse drug reaction | 218
Not completed — Lack of Efficacy | 663
Not completed — Clinical remission | 37
Not completed — Other reasons | 260

BASELINE CHARACTERISTICS:
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4208
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data was available for 4147 participants
  years | 54.6 (13.2)
Gender [Number; unit: participants] — Gender data available for 4157 participants
  participants
    Female | 3199
    Male | 958
Region of Enrollment [Number; unit: participants]
  Germany | 4208

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score (DAS) 28
Description: The Disease Activity Score 28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 score. If the ESR value is missing, the C-reactive protein (CRP) value can be substituted. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set (FAS). Participants with inadequate data or who met other exclusion criteria were not included in the FAS. "n" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
units on a scale
  Month 3 (n=2620) | -1.5 (1.3)
  Month 6 (n=2243 | -1.8 (1.4)
  Month 9 (n=1877) | -1.9 (1.4)
  Month 12 (n=1776) | -2.0 (1.4)
  Month 18 (n=1519) | -2.1 (1.4)
  Month 24 (n=1248) | -2.2 (1.4)

2. Primary Outcome: Percentage of Participants in DAS28 Remission
Description: Clinical remission is defined as a disease activity score (DAS) 28 score of < 2.6. The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (assessed on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28. If the ESR value is missing, the C-reactive protein (CRP) value can be substituted. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity.
Time Frame: Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
percentage of participants
  Month 3 (n=2620) | 18.1
  Month 6 (n=2243) | 22.0
  Month 9 (n=1877) | 26.1
  Month 12 (n=1776) | 27.2
  Month 18 (n=1519) | 29.8
  Month 24 (n=1248) | 34.6

3. Secondary Outcome: Percentage of Participants With a Significant Therapeutic Response
Description: Significant therapeutic response was determined by DAS28 critical difference (Dcrit). A Dcrit response is a statistically determined value that exceeds the threshold of random fluctuation and signifies a positive individual response during treatment. A DAS28-Dcrit individual therapeutic response is defined as a decrease (improvement) in DAS28 from Baseline of ≥ 1.8.
  The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (assessed on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28. If the ESR value is missing, the C-reactive protein (CRP) value can be substituted. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
percentage of participants
  Month 3 (n=2620) | 38.9
  Month 6 (n=2243) | 49.1
  Month 9 (n=1877) | 54.7
  Month 12 (n=1776) | 56.3
  Month 18 (n=1519) | 60.1
  Month 24 (n=1248) | 61.9

4. Secondary Outcome: Percentage of Participants With Low, Moderate and High Disease Activity
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (assessed on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28. If the ESR value is missing, the C-reactive protein (CRP) value can be substituted. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity.
  Low disease activity is defined as a DAS28 score ≤ 3.2; Moderate disease activity as a DAS28 >3.2 to ≤5.1; High disease activity as a DAS28 >5.1.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point
Measure: Number; unit: percentage of participants
Groups:
- Month 0: Baseline
- Month 3: 3 months after inclusion
- Month 6: 6 months after inclusion
- Month 9: 9 months after inclusion
- Month 12: 12 months after inclusion
- Month 18: 18 months after inclusion
- Month 24: 24 months after inclusion
Arm/Group | Month 0 | Month 3 | Month 6 | Month 9 | Month 12 | Month 18 | Month 24
Number analyzed (Participants) | 2950 | 2620 | 2243 | 1877 | 1776 | 1519 | 1248
percentage of participants
  Low disease activity | 0.0 | 30.2 | 36.5 | 41.8 | 43.7 | 46.7 | 51.4
  Moderate disease ctivity | 35.7 | 45.9 | 45.6 | 43.9 | 43.1 | 41.7 | 37.7
  High disease activity | 64.3 | 23.9 | 17.9 | 14.3 | 13.2 | 11.6 | 10.9

5. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Over Time
Description: Erythrocyte sedimentation rate (ESR) indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
mm/hour
  Month 0 (n=2900) | 32.1 (22.0)
  Month 3 (n=2684) | 23.2 (20.2)
  Month 6 (n=2259) | 22.1 (19.1)
  Month 9 (n=1910) | 21.6 (18.2)
  Month 12 (n=1805) | 21.4 (17.9)
  Month 18 (n=1515) | 21.0 (17.5)
  Month 24 (n=1263) | 21.2 (18.7)

6. Secondary Outcome: C-Reactive Protein (CRP) Levels Over Time
Description: C-Reactive Protein (CRP) was measured from blood samples as a marker for inflammation. Higher levels are indicative of more inflammation. Normal concentration in healthy human serum is usually lower than 10 mg/L, slightly increasing with age.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
mg/L
  Month 0 (n=2899) | 20.0 (36.6)
  Month 3 (n=2677) | 11.9 (31.9)
  Month 6 (n=2289) | 9.2 (19.5)
  Month 9 (n=1936) | 8.1 (15.8)
  Month 12 (n=1813) | 8.0 (17.7)
  Month 18 (n=1537) | 6.6 (11.9)
  Month 24 (n=1297) | 5.7 (10.9)

7. Secondary Outcome: Tender Joint Count (TJC) Over Time
Description: Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
tender joints
  Month 0 (n=2950) | 10.6 (6.7)
  Month 3 (n=2778) | 5.4 (6.1)
  Month 6 (n=2393) | 4.3 (5.4)
  Month 9 (n=2010) | 3.9 (5.4)
  Month 12 (n=1886) | 3.6 (5.0)
  Month 18 (n=1621) | 3.4 (4.9)
  Month 24 (n=1339) | 3.1 (4.5)

8. Secondary Outcome: Swollen Joint Count (SJC) Over Time
Description: Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
swollen joints
  Month 0 (n=2950) | 7.7 (5.6)
  Month 3 (n=2768) | 3.7 (4.6)
  Month 6 (n=2375) | 3.0 (4.1)
  Month 9 (n=2003) | 2.6 (3.8)
  Month 12 (n=1868) | 2.4 (3.7)
  Month 18 (n=1609) | 2.1 (3.4)
  Month 24 (n=1326) | 2.0 (3.4)

9. Secondary Outcome: Hannover Functional Questionnaire (FFbH) Over Time
Description: A self-administered patient questionnaire used to assess patient function based on 18 questions. The numerically coded responses to the questions are added to provide a total patient score. The FFbH was calculated from this patient score by the following formula:
  FFbH = (patient score x 100) ÷ 2 (number of valid responses). The resulting FFbH score reflects the degree of remaining functional capacity where 0 indicates maximal impairment and 100 indicates maximal functional capacity.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
units on a scale
  Month 0 (n=2938) | 61.9 (22.4)
  Month 3 (n=2755) | 68.4 (22.5)
  Month 6 (n=2369) | 70.4 (22.2)
  Month 9 (n=1997) | 71.3 (22.5)
  Month 12 (n=1882) | 71.9 (22.4)
  Month 18 (n=1623) | 72.4 (22.5)
  Month 24 (n=1341) | 72.7 (22.7)

10. Secondary Outcome: Patients Global Assessment of Disease Activity Over Time
Description: Participants indicated their global assessment of disease activity over the last 7 days on a visual analog scale (VAS) from 0 (best) to 10 (worst) cm; lower scores indicate better patient status.
Time Frame: Baseline and Months 3, 6, 9, 12, 18 and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
cm
  Month 0 (n=2950) | 6.3 (1.9)
  Month 3 (n=2731) | 4.7 (2.2)
  Month 6 (n=2353) | 4.4 (2.1)
  Month 9 (n=1975) | 4.2 (2.1)
  Month 12 (n=1869) | 4.1 (2.1)
  Month 18 (n=1609) | 4.0 (2.1)
  Month 24 (n=1339) | 3.8 (2.1)

11. Secondary Outcome: Participants Assessment of Fatigue Over Time
Description: Participants indicated their level of fatigue over the last 7 days on a visual analog scale (VAS) from 0 (best) to 10 (worst) cm; lower scores indicate better patient status.
Time Frame: Baseline and Month 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
cm
  Month 0 (n=2940) | 5.8 (2.5)
  Month 3 (n=2727) | 4.5 (2.7)
  Month 6 (n=2351) | 4.2 (2.6)
  Month 9 (n=1976) | 4.0 (2.6)
  Month 12 (n=1864) | 4.0 (2.6)
  Month 18 (n=1608) | 3.9 (2.6)
  Month 24 (n=1335) | 3.7 (2.6)

12. Secondary Outcome: Participants Assessment of Pain Over Time
Description: Participants indicated their level of pain over the last 7 days on a visual analog scale (VAS) from 0 (best) to 10 (worst) cm; lower scores indicate better patient status.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
cm
  Month 0 (n=2942) | 6.4 (2.1)
  Month 3 (n=2732) | 4.5 (2.4)
  Month 6 (n=2356) | 4.2 (2.4)
  Month 9 (n=1973) | 4.1 (2.4)
  Month 12 (n=1866) | 3.9 (2.4)
  Month 18 (n=1609) | 3.9 (2.4)
  Month 24 (n=1339) | 3.7 (2.4)

13. Secondary Outcome: Percentage of Participants With Impairment in Daily Activities
Description: Participants were asked to report how many days of impairment in daily activities they had experienced in the last 4 weeks.
Time Frame: Baseline and Months 3, 6, 9, 18, and 24
Population: Full analysis set with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Month 0 | Month 3 | Month 6 | Month 9 | Month 18 | Month 24
Number analyzed (Participants) | 2864 | 2648 | 2288 | 1914 | 1513 | 1302
percentage of participants
  No days of impairment | 19.7 | 35.8 | 40.3 | 45.7 | 51.4 | 52.1
  Less than 7 days of impairment | 28.5 | 36.3 | 35.5 | 33.3 | 30.0 | 30.4
  7 to 14 days of impairment | 28.8 | 16.1 | 14.9 | 13.2 | 12.0 | 10.8
  More than 14 days of impairment | 23.0 | 11.7 | 9.4 | 7.8 | 6.7 | 6.7

14. Secondary Outcome: Number of Days Missed From Work Due to Rheumatoid Arthritis
Description: Participants reported the number of days they had missed from work in the prior 6 months. The Baseline measurement includes data for the prior 12 months.
Time Frame: Baseline and Months 6, 12, 18, and 24
Population: Full analysis set participants who were employed and with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
days
  Month 0 (n=1168) | 20.6 (52.4)
  Month 6 (n=938) | 9.9 (33.2)
  Month 12 (n=728) | 4.4 (21.3)
  Month 18 (n=604) | 5.2 (27.1)
  Month 24 (n=507) | 3.8 (17.9)

15. Secondary Outcome: Percentage of Participants With In-patient Hospitalization
Description: The percentage of participants with in-patient hospitalization in the prior 6 months. Baseline data includes in-patient hospitalizations that occurred within the prior 12 months.
Time Frame: Month 6, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 2950
percentage of participants
  Baseline (n=2893) | 21.6
  Month 6 (n=2293) | 7.2
  Month 12 (n=1844) | 5.8
  Month 18 (n=1584) | 5.4
  Month 24 (n=1320) | 3.6

16. Secondary Outcome: Percentage of Participants on Concomitant Rheumatoid Arthritis and Pain Relief/Anti-inflammatory Medication
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Full analysis set with available data at each time point (indicated by n)
Measure: Number; unit: percentage of participants
Arm/Group | Month 0 | Month 3 | Month 6 | Month 9 | Month 12 | Month 18 | Month 24
Number analyzed (Participants) | 2950 | 2820 | 2415 | 2041 | 1917 | 1651 | 1372
percentage of participants
  Methotrexate | 54.0 | 52.3 | 53.2 | 53.1 | 53.2 | 52.9 | 51.0
  Sulfasalazine | 6.2 | 3.7 | 3.6 | 3.2 | 3.5 | 3.3 | 2.8
  Hydroxychloroquine/Chloroquine | 2.5 | 2.0 | 1.6 | 1.2 | 1.2 | 1.3 | 1.4
  Leflunomide | 22.1 | 18.0 | 15.9 | 15.3 | 15.0 | 14.1 | 12.7
  Other disease-modifying antirheumatic drug | 4.5 | 2.8 | 2.5 | 2.3 | 2.0 | 2.2 | 2.1
  Analgesics | 21.8 | 15.4 | 14.9 | 14.0 | 12.9 | 11.7 | 12.0
  Non-steroidal anti-inflammatory drug | 46.1 | 36.9 | 34.2 | 33.9 | 32.7 | 31.7 | 30.5
  Cyclo-oxygenase 2 (COX-2) Inhibitors | 12.4 | 10.4 | 10.2 | 9.6 | 9.2 | 9.6 | 9.7
  Systemic glucocorticoids | 80.9 | 73.4 | 69.1 | 65.7 | 62.1 | 58.8 | 57.4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected throughout the 24-month period.
Description: During this non-interventional study, clinicians were asked to report AEs considered to be related to the study medication for all patients who received at least one dose of adalimumab (safety set; N = 4208).
Arm/Group | Rheumatoid Arthritis
Serious Adverse Events (participants affected / at risk) | 245/4208
Other Adverse Events (participants affected / at risk) | 0/4208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (N=4208)
Nasopharyngitis (Infections and infestations) | 11
Pneumonia (Infections and infestations) | 10
Bronchitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 4
Bronchopneumonia (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Laryngitis (Infections and infestations) | 3
Rash pustular (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Gastrointestinal infection (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Localized infection (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Device-related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Encephalitis viral (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Infection susceptibility increased (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyothorax (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Infection site erythema (General disorders) | 11
Injection site pruritus (General disorders) | 9
Injection site reaction (General disorders) | 5
Unevaluable event (General disorders) | 5
Pyrexia (General disorders) | 4
Injection site pain (General disorders) | 3
Edema (General disorders) | 2
Fatigue (General disorders) | 2
Inflammation (General disorders) | 2
Injection site swelling (General disorders) | 2
Injection site urticaria (General disorders) | 2
Adverse drug reaction (General disorders) | 1
Chills (General disorders) | 1
Condition aggravated (General disorders) | 1
Death (General disorders) | 1
Disease recurrence (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site scab (General disorders) | 1
Local swelling (General disorders) | 1
Malaise (General disorders) | 1
Mucosal dryness (General disorders) | 1
Obstruction (General disorders) | 1
Peripheral edema (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 3
Pruritus generalized (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Skin discomfort (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Hypoesthesia oral (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Mouth edema (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Tongue blistering (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Hospitalization (Surgical and medical procedures) | 6
Joint arthroplasty (Surgical and medical procedures) | 4
Synovectomy (Surgical and medical procedures) | 3
Injection (Surgical and medical procedures) | 2
Surgery (Surgical and medical procedures) | 2
Antibiotic therapy (Surgical and medical procedures) | 1
Arthrodesis (Surgical and medical procedures) | 1
Esophageal operation (Surgical and medical procedures) | 1
Mastoid operation (Surgical and medical procedures) | 1
Mastoidectomy (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Sinus operation (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Therapy cessation (Surgical and medical procedures) | 1
Vertebroplasty (Surgical and medical procedures) | 1
Dizziness (Nervous system disorders) | 6
Cerebrovascular accident (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 3
Anosmia (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hypogeusia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 2
Congestive cardiomyopathy (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 3
Foot fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Bloody airway discharge (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Wound secretion (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary tumor of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urteric cancer local (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Eyelid edema (Eye disorders) | 3
Cataract (Eye disorders) | 1
Eyelid exfoliation (Eye disorders) | 1
Eyelids pruritus (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Arthroscopy (Investigations) | 2
Antinuclar antibody positive (Investigations) | 1
Arteriogram coronary (Investigations) | 1
DNA antibody positive (Investigations) | 1
Electrophoresis protein abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Transaminase increased (Investigations) | 1
Anxiety (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Panic reaction (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Bladder tamponade (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Cystitis hemorrhagic (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nephritis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 3
Flushing (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Anemia hemolytic autoimmune (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.